CLINICAL TRIAL: NCT00001153
Title: Visual Function and Ocular Pigmentation in Albinism
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 760207; 76-EI-0207
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Albinism; Albinism, Ocular; Albinism, Oculocutaneous
Keywords: Albinism; Ocular Albinism; Oculocutaneous Albinism; Tyrosinase Negative; Tyrosinase Positive
MeSH Terms: conditions — Albinism; Albinism, Ocular; Albinism, Oculocutaneous

SUMMARY:
To study the relationship between visual function and ocular (iris, retina/choroidal) pigmentation in patients with albinism and other hypomelanotic disorders. To identify the carrier state in relatives of patients with ocular albinism.

DETAILED DESCRIPTION:
Visual function and ocular pigmentation are being studied in patients with albinism and other disorders associated with hypopigmentation. The degree of ocular pigmentation is assessed clinically by estimating the melanin content of the iris, retinal pigment epithelium, and choroid. Visual function is measured in the conventional manner to study central vision, and electrophysiological methods to detect a misrouting of the visual pathways. The purpose of this study is to document the visual deficit and the pigmentary changes of patients with albinism, to observe their natural course, and to determine whether misrouting of the visual pathways is present and is correlated with pigmentation.

ELIGIBILITY:
Patients have been recruited into the study by referral from an ophthalmologist or pediatrician.

Entrance into the study was dependent upon clinical evidence of decreased or absent pigmentation in skin, hair, and/or eyes.

The definition was purposefully broad to include the broad range of phenotype variations and clinical heterogeneity.

The purpose of the study id to be able to document iris and retina/choroidal pigmentation and correlated these finding with visual function.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 1976-06; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Apkarian P, Shallo-Hoffmann J. VEP projections in congenital nystagmus; VEP asymmetry in albinism: a comparison study. Invest Ophthalmol Vis Sci. 1991 Aug;32(9):2653-61. PMID 1651299
- [Background] Bouzas EA, Caruso RC, Drews-Bankiewicz MA, Kaiser-Kupfer MI. Evoked potential analysis of visual pathways in human albinism. Ophthalmology. 1994 Feb;101(2):309-14. doi: 10.1016/s0161-6420(13)31336-0. PMID 8115151